CLINICAL TRIAL: NCT04796428
Title: Intraclass Safety and Efficacy Comparison Among SGLT-2 Inhibitors in Elderly Patients With Type 2 Diabetes. A Pragmatic, Phase IV, Multicenter, Open-label, Randomised Controlled Trial.
Brief Title: GliflOzin in eLderly Diabetic patiENts: A praGmatic Intraclass Evaluation Trial
Acronym: GOLDEN-AGE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center for Outcomes Research and Clinical Epidemiology, Italy (Other)
Collaborators: Italian Society of Diabetology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRS-2019-00002051
Record Dates: First submitted 2021-03-01; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; dapagliflozin; empagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- canagliflozin (Active Comparator): 100 mg (or 50/850 mg and 50/1000 mg of the fixed association with metformin) or 300 mg (or the 150/850 mg and the 150/1000 mg fixed association with metformin).
  Interventions: Drug: Canagliflozin
- dapagliflozin (Active Comparator): 10 mg (or 5/850 mg and 5/1000 mg of the fixed association with metformin; or 10/5 mg of the fixed dapagliflozin / saxagliptin combination)
  Interventions: Drug: Dapagliflozin
- empagliflozin (Active Comparator): 10 mg (or 5/850 mg and 5/1000 mg of the fixed association with metformin; or 5/5 mg of the empagliflozin / linagliptin combination) or 25 mg (or the 12.5/850 mg and the 12.5/1000 mg fixed association with metformin; or the 12.5/5 mg empagliflozin / linagliptin combination).
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Canagliflozin — Canagliflozin If the patient is already on metformin, the fixed combination Canagliflozin / Metformin can be used.
  Arms: canagliflozin
Drug: Dapagliflozin — Dapagliflozin If the patient is already on metformin, the fixed combination dapagliflozin / metformin can be used.
  If the patient is already on a DPP-4 inhibitor, the fixed dose combination dapagliflozin / saxagliptin can be used.
  Arms: dapagliflozin
Drug: Empagliflozin — If the patient is already on metformin, the fixed combination empagliflozin / metformin can be used.
  If the patient is already on a DPP-4 inhibitor, the fixed dose combination empagliflozin / linagliptin can be used.
  Arms: empagliflozin

SUMMARY:
Three SGLT2i were commercially available in Italy at the time the trial was designed: canagliflozin, dapagliflozin, and empagliflozin. Preliminary evidence suggests that the higher dose canagliflozin (300 mg/day) might exert a stronger glucose-lowering effect than dapagliflozin or empagliflozin. The clinical relevance of this putative difference is however unknown. On the other side, the use of canagliflozin, but not empagliflozin and dapagliflozin, has been associated with an increased risk of some adverse events, namely bone fractures and lower limb amputations. Currently, the available information on the efficacy and safety of SGLT2i in elderly (70+ years) patients with type 2 diabetes are is very scant. Thus, a compelling need now exists of comparing efficacy and safety of the commercially available SGLT2i in a population of frail patients at high risk of cardiovascular and renal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age 70+ years
* Male or female
* Prevalent cardiovascular disease (symptomatic or asymptomatic) or eGFR <90 ml/min/1.73 m2 and above the lower limit for initiation of SGLT2i according to label (currently eGFR <60 ml/min/1.73 m2)
* HbA1c above individualized target
* Indication to add SGLT2i

Exclusion Criteria:

* Age >90 years
* Estimated life expectancy <1 year
* Very high risk of genitourinary tract infections (>2 events in the last 6 months)
* Recent weight loss (>5% in <6 months)
* Inability to provide informed consent

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1167 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Up to 24 months
  The primary objective is to compare the proportion of patients treated with each SGLT2i drug, who achieve the individualized HbA1c target without level-2 hypoglycaemia.

SECONDARY OUTCOMES:
Secondary Objectives - HbA1c | Up to 24 months
  Change in HbA1c level (as a continuous variable) - %
Secondary Objectives - body weight | Up to 24 months
  Change in body weight (as a continuous variable) - Kg
Secondary Objectives - systolic blood pressure | Up to 24 months
  Change in systolic blood pressure (as a continuous variable) - mmHG
Secondary Objectives - e-GFR | Up to 24 months
  Change in e-GFR (as a continuous variable). The slope of eGFR decline will be calculated over time in the three treated groups - mL/min
Secondary Objectives - urinary albumin excretion rate | Up to 24 months
  Change in urinary albumin excretion rate (as a continuous variable) - mg/L
Secondary Objectives - medications | Up to 24 months
  Change concomitant medications and their daily dosages
Secondary Objectives - treatment satisfaction | Up to 24 months
  Change in treatment satisfaction quantified as Diabetes Treatment Satisfaction Questionnaire (DTSQ).
Secondary Objectives - biomarkers | Up to 24 months
  Plasma/serum biomarkers of bone metabolism and cardiac function (in a subset of patients) with physiological parameter

OTHER OUTCOMES:
Safety Objectives | Up to 24 months
  Hospitalization for any cause
Safety Objectives | Up to 24 months
  Hospitalization for heart failure and/or cardiovascular causes
Safety Objectives | Up to 24 months
  All-cause death and Cardiovascular death
Safety Objectives | Up to 24 months
  Severe hypoglycemia
Safety Objectives | Up to 24 months
  Genitourinary tract infections
Safety Objectives | Up to 24 months
  Dehydration / hypovolemia events
Safety Objectives | Up to 24 months
  Bone fractures
Safety Objectives | Up to 24 months
  Leg/foot amputations
Safety Objectives | Up to 24 months
  Diabetic ketoacidosis

IPD SHARING:
Plan to Share IPD: No